CLINICAL TRIAL: NCT06702748
Title: Research on New Technologies for the Diagnosis and Treatment of Cardiovascular Diseases-Multi-parameter Noninvasive Early Diagnosis of Coronary Microvascular Diseases Series I: Clinical Study Protocol for a New Method of Evaluating Coronary Microvessels Based on Coronary IMR Calculated from Coronary Angiography Images
Brief Title: Prognostic Values of Coronary Microvascular Dysfunction Patients Treated with Rotational Atherectomy During Percutaneous Coronary Intervention
Status: Active, not recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 20220940-3
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Coronary Arterial Disease (CAD); Coronary Microvascular Dysfunction (CMD)
Keywords: Coronary Microvascular Dysfunction; Index of Microcirculatory Resistance; Coronary artery disease; rotational atherectomy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Coronary microvascular dysfunction: angio-IMR>=25
- Non-Coronary microvascular dysfunction: Angio-IMR<25

SUMMARY:
The goal of this observational study is to learn about the long-term prognostic of coronary microvascular dysfuction in Patients Treated with Rotational Atherectomy During Percutaneous Coronary Intervention.

The main question it aims to answer is: Does the coronary microvascular dysfunction impact the outcomes in Patients Treated with Rotational Atherectomy During Percutaneous Coronary Intervention.

Participants will answer survey questions about their clinical outcomes for 2 years by telephone.

DETAILED DESCRIPTION:
This study was a retrospective, multicenter observational investigation and approved by the local Human Research Ethics Committee and conducted in accordance with the principles outlined in the Helsinki Declaration.Patients aged 18 years or older who had severe coronary calcification and underwent successful RA during PCI were eligible for inclusion in the study. Exclusion criteria included target vessel was chronic total occlusion, poor angiographic image quality, failed RA and RA not used for severe coronary calcification.

Angiography-derived index of microcirculatory resistance was measured in the target vessel treated with RA pre-PCI and post-PCI and blinded and performed by an independent core laboratory.The follow-up entailed the utilization of a multipronged approach, encompassing clinic visits, medical record reviews and telephone contacts.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older who had severe coronary calcification and underwent successful RA during PCI

Exclusion Criteria:

* target vessel was chronic total occlusion, poor angiographic image quality, failed RA and RA not used for severe coronary calcification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who had severe coronary calcification and underwent successful RA during PCI
Sampling Method: Non-Probability Sample
Enrollment: 452 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiac events | 24 months after PCI
  the composite of cardiac death, myocardial reinfarction, target vessel revascularization, and readmission for unstable angina

SECONDARY OUTCOMES:
target vessel failure | 24 months after PCI
  composed of cardiac death, target vessel myocardial infarction, target vessel revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- 88 Jiefang Road, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
undecided